CLINICAL TRIAL: NCT00254878
Title: A 7 Week Multicenter, Double-Blind, Randomized, Placebo-Controlled Cross-Over Evaluation of the Efficacy and Safety of Two Different Brands of Modified-Release Oral Dosage Forms of Methylphenidate-HCl (20 mg, q.d.) in Children With Attention Deficit Hyperactivity Disorder (ADHD) Aged 6 - 14
Brief Title: Placebo-Controlled Comparison of Two Different Brands of Modified-Release Oral Dosage Forms Regarding Safety and Efficacy in Children With Attention Deficit Hyperactivity Disorder (ADHD) Aged 6 - 14
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRIT124DDE01
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: ADHD
Keywords: ADHD, Methylphenidate hydrochloride, modified-release
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate hydrochloride

SUMMARY:
Currently two different brands of modified-release formulations are providing 50% immediate release beads/pellets and 50% extended release beads/pellets, resulting in a rapid onset and dual peak concentrations of plasma methylphenidate. One is manufactured by Novartis, the other one by Medice (Germany).

The objective of the study is to test the hypothesis that the Novartis product is superior to placebo and is clinically not inferior to the formulation manufactured by Medice.

DETAILED DESCRIPTION:
Currently two different brands of modified-release formulations are providing 50% immediate release beads/pellets and 50% extended release beads/pellets, resulting in a rapid onset and dual peak concentrations of plasma methylphenidate. One is manufactured by Novartis, the other one by Medice (Germany).

The objective of the study is to test the hypothesis that the Novartis product is superior to placebo and is clinically not inferior to the formulation manufactured by Medice.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following inclusion criteria will be eligible for enrollment in the study:

* Male and female patients aged 6-14.
* Patients having a diagnosis of ADHD of any type according to DSM-IV criteria, as established by history, psychiatric examination and a structured diagnostic interview (Kiddie-Sads-Present and Lifetime Version)
* Patients, whose symptoms are adequately controlled by a stable and well-tolerated dose of a immediate release methylphenidate equivalent of 20mg for one month before screening.

Exclusion Criteria:

* Patients with comorbid psychiatric conditions with symptoms requiring current pharmacological treatment (e.g. major depression, psychosis).
* Patients who are taking any concomitant medications likely to interfere with the study drug or confound efficacy or safety assessments, e.g.

  * Tricyclic antidepressants, buproprion, clonidine, buspirone 2 weeks before randomization.
  * Atomoxetine 2 weeks before randomization.
  * Fluoxetine or antipsychotics 1 month before randomization.
  * Pemoline and amphetamines 1 week before randomization.
* Patients with a known non-response to methylphenidate.

Other protocol-defined exclusion criteria may apply.

Ages: 6 Years to 14 Years | Sex: All
Age Groups: Child
Enrollment: 130
Dates: Start 2005-10; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Attention and deportment measured at 1.5, 3.0 and 4.5 hours after drug intake

SECONDARY OUTCOMES:
7 week's treatment with two different brands of modified-release oral dosage forms of methylphenidate-HCl on attention, deportment, behavior and math in children with attention deficit hyperactivity disorder (ADHD) aged 6 - 14
Safety of 7 week's treatment with two different brands of modified-release oral dosage forms of methylphenidate-HCl

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, Freiburg im Breisgau, Germany